CLINICAL TRIAL: NCT00773019
Title: SynchroMed II Programmable Drug Infusion System Post-Approval Study
Brief Title: SynchroMed II Post-Approval Study
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1607
Record Dates: First submitted 2008-08-21; First posted 2008-10-16 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Severe Spasticity; Chronic Pain
Keywords: infusion pump; implantable; performance
MeSH Terms: conditions — Muscle Spasticity; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Refills (SynchroMed® II Programmable Drug Infusion Pump) — Refill information at 1, 6, and 12 months post-implant, as well as any additional refills required from implant through end of study. Amount removed from the pump (taken from syringe), Amount placed in the pump (from syringe),Pump predicted amount remaining in the pump.

SUMMARY:
This FDA Condition of Approval study will include up to 100 subjects at up to 13 US centers. Subjects are selected from those evaluated and planning to receive a SynchroMed II drug infusion system for treatment of severe spasticity or chronic pain. Subjects must return for refill visits at 1, 6, and 12 months. In addition, subjects return for any other medically necessary refills. Information is collected on all refills and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic intractable severe spasticity or chronic pain requiring intrathecal delivery of medication
* Have undergone a pre-implant assessment and determined to be an appropriate candidate for implantation of an infusion system
* Be geographically stable and willing to return to the study center for follow-up visits
* Subject, or subject's legal representative, has signed informed consent form prior to any study-related procedures
* Age is at least 18 years of age at time of enrollment

Exclusion Criteria:

* Have a condition in which the pump cannot be implanted 2.5 cm or less from the surface of the skin
* Have an ongoing infection prior to implant
* Have insufficient body mass to accept the pump bulk and weight
* Are unable or unwilling to adhere to the study protocol
* Have an estimated life expectancy of less than twelve months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects planning to receive a new or replacement drug pump.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Compare the observed volume of drug dispensed by the pump to the programmer's calculated volume of drug dispensed | six months

SECONDARY OUTCOMES:
Characterize adverse events experienced with the drug infusion system | one year